CLINICAL TRIAL: NCT02801955
Title: Predictive Value of Serum and Peritoneal CEA and CA 19-9 for TNM Stage and Peritoneal Dissemination of Gastric Adenocarcinoma
Brief Title: Serum and Peritoneal CEA and CA 19-9 for Gastric Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Mustafa Hasbahceci, Associate Professor of General Surgery, Bezmialem Vakif University
Other Study IDs: GastCancTmMark2016
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Gastric Adenocarcinoma
Keywords: gastric adenocarcinoma; tumor markers; peritoneal cytology
MeSH Terms: interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tumor marker: serum CEA and CA 19-9 levels in patients with curative gastrectomy preoperatively and peritoneal CEA and CA 19-9 levels in patients taken at the beginning of curative gastrectomy via sampling of peritoneal washing aspirate
  Interventions: Procedure: gastrectomy; Procedure: sampling of peritoneal washing aspirate

INTERVENTIONS:
Procedure: gastrectomy — radical total/subtotal gastrectomy with D2 lymph node dissection
Procedure: sampling of peritoneal washing aspirate — After thoroughly examination of the peritoneal cavity revealing the absence of peritoneal dissemination, the peritoneal cavity was washed with 200 ml of saline, and at least one third was aspirated from several regions of the peritoneal cavity, including near the primary tumor, the left and right subphrenic areas and the pouch of Douglas with suction tubes to a clean bottle and designated as the peritoneal sample for determination of peritoneal levels of CEA and CA 19-9.

SUMMARY:
For preoperative staging and prediction of peritoneal dissemination of gastric adenocarcinoma, usage of serum and peritoneal levels of carcinoembryonic antigen (CEA) and CA 19-9 may be helpful. Additionally, the prognosis of the patients with gastric adenocarcinoma treated with gastrectrectomy may be associated with serum and peritoneal levels of tumor markers.

DETAILED DESCRIPTION:
Clinical usage of tumor markers on preoperative staging and prediction of peritoneal dissemination of gastric adenocarcinoma is a controversial issue. It has been thought that there is a positive correlation between serum and peritoneal levels of carcinoembryonic antigen (CEA) and CA 19-9 and pathologic features of gastric tumors and peritoneal dissemination.

In this study, it was aimed to evaluate the effect of serum and peritoneal CEA and CA 19-9 to predict TNM stages and peritoneal washing cytology in patients with gastric adenocarcinoma after curative gastrectomy, and to determine predictive value of these measurements to the development of recurrence and death.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically proven gastric adenocarcinoma
* Standard gastrectomy and a D2 lymph node dissection;
* Desire to attend the study protocol

Exclusion Criteria:

* Metastatic or overt peritoneal disseminated cancer
* Undesired reaction to attend the study protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric adenocarcinoma treated with curative gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
TNM stage | through pathologic report completion, an average of 1 month
  TNM stage based on the 7th American Joint Committee on Cancer/International Union Against Cancer tumor, node, metastasis system.

SECONDARY OUTCOMES:
peritoneal washing cytology | through pathologic report completion, an average of 1 month
  detection of positive free peritoneal gastric adenocarcinoma cells.
recurrence/death | through follow-up period, an average of 24 months
  detection of recurrence or development of death

CONTACTS AND LOCATIONS:
Overall Officials: mustafa hasbahceci, assoc. prof., Principal Investigator — bezmialem vakif university faculty of medicine
Locations (1):
- Mustafa Hasbahceci, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No